CLINICAL TRIAL: NCT06461104
Title: Physical Activity in People With Borderline Personality Disorder (PABORD): a Study Protocol for a Pilot Randomised Controlled Trial (RCT)
Brief Title: Physical Activity in People With Borderline Personality Disorder (PABORD)
Acronym: PABORD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1A1B2O3R5D8
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Borderline Personality Disorder
Keywords: Physical Activity; Borderline Personality Disorder; ESM; Females; Global Functioning; Accelerometer; Motivation; Premenstrual Syndrome; Outpatients
MeSH Terms: conditions — Borderline Personality Disorder; Motor Activity; Premenstrual Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This randomised controlled trial (RCT) is designed to evaluate the efficacy of a structured physical activity (PA) programme compared to a psychoeducational intervention on healthy lifestyle in female outpatients aged 18 to 40 years with a diagnosis of Borderline Personality Disorder (BPD). Participants will be randomly assigned to one of two groups: an intervention group that engages in a 12-week structured PA programme preceded by three psychoeducational sessions focused on nutrition, and a control group that receives a 12-week psychoeducational programme on nutrition and PA. The study aims to assess changes in clinical symptoms, PA-related parameters, and various physical, psychological, and biological outcomes at baseline, mid-treatment, end of treatment, and at a 3-month follow-up. This RCT adheres to the Declaration of Helsinki and involves comprehensive informed consent and data processing protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will engage in a 12-week structured PA programme, preceded by three weekly psychoeducational sessions focused on nutrition. This includes three 60-minute PA sessions per week supervised by a personal trainer.
  Interventions: Behavioral: Structured Physical Activity Programme; Behavioral: Psychoeducational Programme
- Control Group (Active Comparator): Participants will receive a 12-week psychoeducational programme on nutrition and PA. This programme includes 8 sessions divided into modules of 2 or 3 lessons each, covering topics such as the benefits of PA and sports, healthy eating habits, and health risks associated with a sedentary lifestyle. Sessions will be conducted by a dietitian and a clinical psychologist. At the end of the trial, control group participants will be offered the opportunity to participate in the same PA programme as the intervention group at no cost.
  Interventions: Behavioral: Psychoeducational Programme

INTERVENTIONS:
Behavioral: Structured Physical Activity Programme — A somatic examination will also be conducted by a sports physician, which will include the assessment of muscle strength, cardiorespiratory fitness, walking gait, blood pressure, and body mass index (BMI). Based on this evaluation, the sports physician will design a personalised physical activity programme for the participants in the intervention group.
  Other Names: Physical Activity
  Arms: Intervention Group
Behavioral: Psychoeducational Programme — The control group undergoes a 12-week psychoeducational programme on nutrition and PA, consisting of 8 sessions. Led by a dietitian and psychologist, topics include PA benefits, healthy eating, and sedentary lifestyle risks. The experimental group receives 3 sessions on dietary habits before starting PA intervention, ensuring differentiation. It's expected the experimental group directly benefits from exercise, while the control group benefits from PA education. At the trial's end, control group members can join the PA programme for free.
  Other Names: Psychoeducation; Psychoeducation Intervention

SUMMARY:
The aim of this Randomised Controlled Trial (RCT) is to test the effects of a structured physical activity (PA) program on symptoms in female outpatients aged 18 to 40 years with a diagnosis of Borderline Personality Disorder (BPD). The main questions it aims to answer are:

1. Does a structured PA program reduce clinical symptoms in patients with BPD?
2. How does the effectiveness of a structured PA program compare to a psychoeducational intervention in reducing clinical symptoms and improving physical activity parameters?

Participants will participate in a 12-week structured PA program preceded by three weekly psychoeducation sessions focused on nutrition (intervention group) or will receive a 12-week psychoeducational program on nutrition and PA (control group).

Researchers will compare the intervention group (structured PA program) and the control group (psychoeducational program) to see if the structured PA program leads to greater improvements in clinical symptoms and physical activity parameters. Moreover, the study includes a multidimensional assessment (physical, psychological, and biological) at four time points: at the start of the treatment (T0), at 6 weeks (mid-treatment, when changes from PA become visible and measurable), at the end of the 3-month treatment period (T3), and at a 3-month follow-up after the treatment (T6).

DETAILED DESCRIPTION:
Background and Objectives This randomised controlled trial (RCT) aims to investigate the effects of a structured physical activity (PA) programme on the symptoms of outpatients who meet DSM-5-TR criteria for Borderline Personality Disorder (BPD). The hypothesis is that these symptoms may improve over the course of the PA treatment. The primary objective is to evaluate the efficacy of a structured PA intervention on reducing clinical symptoms and improving PA-related parameters compared to a psychoeducational intervention on healthy lifestyle.

Study Design The PABORD RCT is a controlled study involving female outpatients aged 18 to 40 years with a BPD diagnosis. Participants will be informed about the study's objectives, procedures, and the potential risks and benefits of the proposed treatments. After confirming inclusion/exclusion criteria, obtaining signed informed consent, and reviewing the data processing information, participants will be randomly assigned to two groups. This trial will be conducted in accordance with the Declaration of Helsinki (World Medical Association, 2013).

Treatment Arms

The study involves two treatment arms:

Intervention Group (n=30): Participants will engage in a 12-week structured PA programme, preceded by three weekly psychoeducational sessions focused on nutrition. This includes three 60-minute PA sessions per week supervised by a personal trainer.

Control Group (n=30): Participants will receive a 12-week psychoeducational programme on nutrition and PA. This programme includes 8 sessions divided into modules of 2 or 3 lessons each, covering topics such as the benefits of PA and sports, healthy eating habits, and health risks associated with a sedentary lifestyle. Sessions will be conducted by a dietitian and a clinical psychologist. At the end of the trial, control group participants will be offered the opportunity to participate in the same PA programme as the intervention group at no cost.

Assessment and Follow-Up

The study includes a multidimensional assessment (physical, psychological, and biological) at four time points: T0 (baseline), 6 weeks (mid-treatment), T3 (end of treatment), and T6 (3-month follow-up). These assessments will include:

* Standardised tests for BPD symptoms and general functioning.
* Physical examinations by a sports physician to create a personalised PA plan and assess health status post-intervention.
* Evaluation of premenstrual syndrome (PMS) and obstetric history to determine potential improvements related to PA.
* Use of an accelerometer for 7 days to monitor movement and sleep-wake patterns, and an app using the Experience Sampling Method (ESM) for real-time mood and psychosocial dimension assessments.
* Use of an app for dietary tracking.
* Blood and saliva sample analysis to detect PA-induced changes at the biological level.

The follow-up aims to determine whether the structured PA intervention results in medium-term improvements in BPD symptoms, sustained PA levels, changes in motivation for PA, and alterations in PMS symptoms. This will be assessed through accelerometer data, ESM mood and social interaction reports, and analysis of selected biomarkers in blood and saliva.

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Age between 18 and 40 years.
* Primary diagnosis of Borderline Personality Disorder (BPD) according to the diagnostic criteria of the DSM-5.
* Outpatient treatment.
* Ability to provide written informed consent.
* Good understanding of the Italian language.
* Proficiency in using a smartphone.
* The presence of ongoing pharmacological and/or psychotherapeutic treatments is not considered an exclusion criterion.

Exclusion Criteria:

* Current pregnancy or planning a pregnancy within the next 6 months.
* Acute psychotic symptoms.
* Comorbidities with Eating Disorders, Substance Use Disorder, and Bipolar Disorder.
* Absolute contraindications to physical exercise, such as medical conditions that interfere with the ability to perform exercise or with the physiological response to exercise tests, e.g., the use of beta-adrenergic blocking agents.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Borderline Personality Disorder Symptomatology | Baseline (start of the study), end of 3-months treatment (week 12), end of 3-months follow-up (week 24)
  The Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) scale measures borderline personality symptomatology. A reduction in score of at least 3.5 indicates improvement, as demonstrated in previous pharmacological treatment studies. Administered at baseline, end of treatment (T3), and end of follow-up (T6) to assess the impact of structured PA treatment on DBP symptomatology. Evaluators blinded to group assignment will obtain and examine outcome measurements.
Improvement of BPD-Related Symptomatology | Baseline (start of the study), end of 3-months treatment (week 12), end of 3-months follow-up (week 24)
  Additional primary outcomes include psychological variables associated with BPD, including sleep hygiene, mood changes, anxiety, impulsivity, and disability impact on daily functioning. Assessment tools include the Experience Sampling Method (ESM), Beck Depression Inventory short form (BDI-13), State-Trait Anxiety Inventory (STAI-Y), Impulsive Behavior Scale (UPPS-P), World Health Organization Disability Assessment Schedule (WHODAS 2.0), and Premenstrual Symptom Screening Tool (PSST). ESM utilizes a custom app for real-time evaluation, while other tools are self-reported questionnaires administered at different time points throughout the study.

SECONDARY OUTCOMES:
Improvement of Physical Activity-Related Parameters | Baseline (start of the study), week 6 (half of the 3-months treatment), end of 3-months treatment (week 12), end of 3-months follow-up (week 24)
  The secondary outcomes aim to measure increased physical activity (PA) intensity and quantity using actigraphic, dynamometric measures, and questionnaires at various intervals. Expected physical health improvements include enhanced muscle strength, cardiorespiratory fitness, blood pressure, and BMI. Biological markers such as BDNF, kynurenine, cortisol, and DHEA, as well as specific biomarkers like agrin and Nf-L, will be analyzed post-PA intervention. Additional assessments cover innovative biomarkers, resting blood glucose, and basic hematological analyses. Motivation and self-regulation will be assessed using validated Italian versions of BREQ-3, P-scale, and RSES.
Reduction of Premenstrual Symptom Exacerbation | Baseline (start of the study), end of 3-months treatment (week 12), end of 3-months follow-up (week 24)
  The presence, severity, and changes in premenstrual symptoms will be assessed using the Premenstrual Symptom Screening Tool (PSST) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Girolamo, MD, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Girolamo G, Leone S, D'Addazio M, Toffol E, Martinelli A, Bellini S, Calza S, Carnevale M, Cattane N, Cattaneo A, Ghidoni R, Longobardi A, Maffezzoni D, Martella D, Meloni S, Mombelli E, Pogliaghi S, Saraceno C, Tura GB, Rossi R. Physical Activity in young female outpatients with BORderline personality Disorder (PABORD): a study protocol for a randomized controlled trial (RCT). Trials. 2024 Oct 16;25(1):685. doi: 10.1186/s13063-024-08525-8. PMID 39415283